CLINICAL TRIAL: NCT03501069
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Oral Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TAK-418 in Healthy Female Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of Single and Multiple Oral Dose of TAK-418 in Healthy Female Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision; no human safety concern; evaluating preclinical toxicology finding
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: TAK-418-1003; U1111-1209-4647 (Other: WHO)
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — TAK-418

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Non-Japanese Cohort 1: TAK-418 120 mg and TAK-418 160 mg (Experimental): TAK-418 120 milligram (mg) or TAK-418 matching placebo, capsule, orally, once on Day 1 of Period A followed by a minimum of 14 days of washout period, followed by TAK-418 160 mg or TAK-418 matching placebo, capsule, orally, once on Day 1 of Period B. The actual TAK-418 dose for Period B will be determined based on safety, tolerability, and PK data available from the previous dose in Period A.
  Interventions: Drug: TAK-418; Drug: TAK-418 Matching Placebo
- Non-Japanese Cohort 2: TAK-418 20 mg (Experimental): TAK-418 20 mg or TAK-418 matching placebo, capsule, orally, once daily for 10 days.
  Interventions: Drug: TAK-418; Drug: TAK-418 Matching Placebo
- Non-Japanese Cohort 3: TAK-418 40 mg (Experimental): TAK-418 40 mg or TAK-418 matching placebo, capsule, orally, once daily for 10 days. The actual TAK-418 dose for Cohort 3 will be determined based on safety, tolerability, and PK data available from the previous doses.
  Interventions: Drug: TAK-418; Drug: TAK-418 Matching Placebo
- Non-Japanese Cohort 4: TAK-418 60 mg (Experimental): TAK-418 60 mg or TAK-418 matching placebo, capsule, orally, once daily for 10 days. The actual TAK-418 dose for Cohort 4 will be determined based on safety, tolerability, and PK data available from the previous doses.
  Interventions: Drug: TAK-418; Drug: TAK-418 Matching Placebo
- Japanese Cohort 5: TAK-418 20 mg (Experimental): TAK-418 20 mg or TAK-418 matching placebo, capsule, orally, once daily for 10 days. The actual TAK-418 dose for Cohort 5 will be determined based on safety, tolerability, and PK data available from the previous doses.
  Interventions: Drug: TAK-418; Drug: TAK-418 Matching Placebo
- Japanese Cohort 6: TAK-418 40 mg (Experimental): TAK-418 40 mg or TAK-418 matching placebo, capsule, orally, once daily for 10 days. The actual TAK-418 dose for Cohort 6 will be determined based on safety, tolerability, and PK data available from the previous doses.
  Interventions: Drug: TAK-418; Drug: TAK-418 Matching Placebo

INTERVENTIONS:
Drug: TAK-418 — TAK-418 capsules.
Drug: TAK-418 Matching Placebo — TAK-418 matching placebo capsules.

SUMMARY:
The purpose of this study is to characterize safety and tolerability of TAK-418 in non-Japanese and Japanese healthy female participants when administered at single or multiple (once daily [QD]) oral doses.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-418. This study will assess the safety, tolerability, PK and PD of single and multiple rising doses of TAK-418 in healthy Japanese or non-Japanese females.

The study will enroll approximately 48 participants in 6 cohorts and each cohort will have 8 participants. The study will include 2 parts: single rising dose (SRD) in Cohort 1 and multiple rising dose (MRD) in Cohorts 2 to 6. Cohort 3 will include cerebrospinal fluid (CSF) collection. Participants will be randomly assigned (by chance, like flipping a coin) to one of the 6 cohorts.

This two-center trial will be conducted in the United States. The overall time to participate in Cohort 1 of this study is approximately 105 days and 98 days in Cohort 2. Participants will be contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has a body mass index (BMI) greater than or equal to (>=) 18.5 and less than or equal to (<=) 30.0 kilogram per square meter (kg/m^2) at the Screening Visit. (Cohorts 1 to 4 only).
2. Is a nonsmoker who has not used tobacco- or nicotine-containing products (example, nicotine patch) for at least 6 months before administration of the first dose of trial drug or invasive procedure.
3. The participant either is of nonchildbearing potential, OR, if of childbearing potential, is using a highly effective method of contraception with low user dependency during the entire duration of the study.

For Cohorts 5 and 6 (Japanese participants) only:

1. Has a BMI >=18.0 and <= 26.0 kg/m^2, at the Screening Visit.

Exclusion Criteria:

1. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), or human immunodeficiency virus (HIV) antibody/antigen, at Screening.
2. Had major surgery, donated or lost 1 unit of blood (approximately 500 milliliter [mL]) within 4 weeks before the Screening Visit.
3. Has a history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce] per day).
4. Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
5. Has a substance abuse disorder.
6. Has risk of suicide according to the investigator's clinical judgment per Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening or has made a suicide attempt in the 6 months before Screening.
7. Has luteinizing hormone (LH), follicle-stimulating hormone (FSH), or estradiol levels that are clinically abnormal.
8. Has a resting heart rate outside of the range of 50 to 100 beats per minute, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1).

For Cohort 3 only (includes CSF sample collection):

1. Has had CSF collection performed within 30 days before Check-in (Day -1).
2. Has significant vertebral deformities (scoliosis or kyphosis) that, in the opinion of the investigator, may interfere with the lumbar puncture procedure.
3. Has a local infection at the puncture site.
4. Has thrombocytopenia or other suspected bleeding tendencies noted before the procedure.
5. Has developed signs and symptoms of spinal radiculopathy, including lower extremity pain and paresthesia.
6. Has any focal neurological deficit that might suggest an increase in intracranial pressure.
7. Has any abnormal finding on ophthalmological assessment/fundoscopy indicative of raised intracranial pressure (that is, optic disc swelling/edema; or [uncontrolled] hypertensive retinopathy).
8. Regularly has moderate-to-severe headaches requiring analgesics.
9. Has any bleeding abnormality or history of bleeding abnormalities.
10. Has abnormal coagulation tests (prothrombin time [PT]/international normalized ratio [INR], partial thromboplastin time [PTT]) at Screening.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Parexel International, Glendale, California
  - PRA Health Sciences, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Yin W, Arkilo D, Khudyakov P, Hazel J, Gupta S, Quinton MS, Lin J, Hartman DS, Bednar MM, Rosen L, Wendland JR. Safety, pharmacokinetics and pharmacodynamics of TAK-418, a novel inhibitor of the epigenetic modulator lysine-specific demethylase 1A. Br J Clin Pharmacol. 2021 Dec;87(12):4756-4768. doi: 10.1111/bcp.14912. Epub 2021 Jun 10. PMID 33990969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 30 May 2018 to 26 December 2018.
Pre-assignment Details: Healthy female participants were enrolled to receive TAK-418 as single rising dose (SRD) dose of 120 milligram (mg), or 160 mg (non-Japanese cohort), and/or placebo in a crossover fashion; and multiple rising dose (MRD) of 20 mg, 60 mg, 160 mg (non-Japanese cohort) or 20 mg (Japanese cohort). The study was terminated early due to business decision.
Groups:
- Non-Japanese Cohort 1: TAK-418 120 mg + Placebo: TAK-418 120 mg capsule, orally, once on Day 1 of Period A, followed by a washout period of at least 14 days, further followed by TAK-418 120 mg placebo-matching capsule, orally, once on Day 1 of Period B.
- Non-Japanese Cohort 1: TAK-418 120 mg + TAK-418 160 mg: TAK-418 120 mg capsule, orally, once on Day 1 of Period A, followed by a washout period of at least 14 days, further followed by TAK-418 160 mg capsule, orally, once on Day 1 of Period B.
- Non-Japanese Cohort 1: Placebo + TAK-418 160 mg: TAK-418 160 mg placebo-matching capsule, orally, once on Day 1 of Period A, followed by a washout period of at least 14 days, further followed by TAK-418 160 mg capsule, orally, once on Day 1 of Period B.
- Non-Japanese Cohorts 2 to 4: Pooled Placebo; Japanese Cohort 5: Placebo: TAK-418 placebo-matching capsule, orally, once daily for 10 days.
- Non-Japanese Cohort 2: TAK-418 20 mg; Japanese Cohort 5: TAK-418 20 mg: TAK-418 20 mg, capsule, orally, once daily for 10 days.
- Non-Japanese Cohort 3: TAK-418 60 mg: TAK-418 60 mg, capsule, orally, once daily for 10 days.
- Non-Japanese Cohort 4: TAK-418 160 mg: TAK-418 160 mg, capsule, orally, once daily for 10 days.
Period: Period A
Arm/Group | Non-Japanese Cohort 1: TAK-418 120 mg + Placebo | Non-Japanese Cohort 1: TAK-418 120 mg + TAK-418 160 mg | Non-Japanese Cohort 1: Placebo + TAK-418 160 mg | Non-Japanese Cohorts 2 to 4: Pooled Placebo | Japanese Cohort 5: Placebo | Non-Japanese Cohort 2: TAK-418 20 mg | Non-Japanese Cohort 3: TAK-418 60 mg | Non-Japanese Cohort 4: TAK-418 160 mg | Japanese Cohort 5: TAK-418 20 mg
Started | 2 | 4 | 2 | 5 | 1 | 6 | 6 | 3 | 3
Completed | 2 | 4 | 2 | 5 | 1 | 6 | 6 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (at Least 14 Days)
Arm/Group | Non-Japanese Cohort 1: TAK-418 120 mg + Placebo | Non-Japanese Cohort 1: TAK-418 120 mg + TAK-418 160 mg | Non-Japanese Cohort 1: Placebo + TAK-418 160 mg | Non-Japanese Cohorts 2 to 4: Pooled Placebo | Japanese Cohort 5: Placebo | Non-Japanese Cohort 2: TAK-418 20 mg | Non-Japanese Cohort 3: TAK-418 60 mg | Non-Japanese Cohort 4: TAK-418 160 mg | Japanese Cohort 5: TAK-418 20 mg
Started | 2 | 4 | 2 | 0 (Participants other than Cohort 1 were not to continue in subsequent Periods after Period A.) | 0 (Participants other than Cohort 1 were not to continue in subsequent Periods after Period A.) | 0 (Participants other than Cohort 1 were not to continue in subsequent Periods after Period A.) | 0 (Participants other than Cohort 1 were not to continue in subsequent Periods after Period A.) | 0 (Participants other than Cohort 1 were not to continue in subsequent Periods after Period A.) | 0 (Participants other than Cohort 1 were not to continue in subsequent Periods after Period A.)
Completed | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period B
Arm/Group | Non-Japanese Cohort 1: TAK-418 120 mg + Placebo | Non-Japanese Cohort 1: TAK-418 120 mg + TAK-418 160 mg | Non-Japanese Cohort 1: Placebo + TAK-418 160 mg | Non-Japanese Cohorts 2 to 4: Pooled Placebo | Japanese Cohort 5: Placebo | Non-Japanese Cohort 2: TAK-418 20 mg | Non-Japanese Cohort 3: TAK-418 60 mg | Non-Japanese Cohort 4: TAK-418 160 mg | Japanese Cohort 5: TAK-418 20 mg
Started | 2 | 4 | 2 | 0 (Participants other than Cohort 1 were not to continue in subsequent Periods after Period A.) | 0 (Participants other than Cohort 1 were not to continue in subsequent Periods after Period A.) | 0 (Participants other than Cohort 1 were not to continue in subsequent Periods after Period A.) | 0 (Participants other than Cohort 1 were not to continue in subsequent Periods after Period A.) | 0 (Participants other than Cohort 1 were not to continue in subsequent Periods after Period A.) | 0 (Participants other than Cohort 1 were not to continue in subsequent Periods after Period A.)
Completed | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Japanese Cohort 1: TAK-418 120 mg + Placebo | Non-Japanese Cohort 1: TAK-418 120 mg + TAK-418 160 mg | Non-Japanese Cohort 1: Placebo + TAK-418 160 mg | Non-Japanese Cohorts 2 to 4: Pooled Placebo | Japanese Cohort 5: Placebo | Non-Japanese Cohort 2: TAK-418 20 mg | Non-Japanese Cohort 3: TAK-418 60 mg | Non-Japanese Cohort 4: TAK-418 160 mg | Japanese Cohort 5: TAK-418 20 mg | Total
Number analyzed (Participants) | 2 | 4 | 2 | 5 | 1 | 6 | 6 | 3 | 3 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (7.78) | 39.8 (11.32) | 39.0 (18.38) | 47.8 (11.78) | 49.0 (NA) — Standard deviation was not estimable since only one participant was analyzed. | 39.2 (12.32) | 46.7 (10.93) | 43.3 (4.04) | 50.3 (3.51) | 43.4 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 5 | 1 | 6 | 6 | 3 | 3 | 32
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 4
  Not Hispanic or Latino | 2 | 3 | 2 | 4 | 1 | 6 | 5 | 2 | 3 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 6
  White | 1 | 3 | 0 | 4 | 0 | 6 | 5 | 3 | 0 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 4 | 2 | 5 | 1 | 6 | 6 | 3 | 3 | 32
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 71.050 (9.8288) | 67.875 (5.5506) | 66.250 (13.7886) | 70.60 (7.090) | 67.90 (NA) — Standard deviation was not estimable since only one participant was analyzed. | 66.60 (6.690) | 70.22 (9.100) | 78.27 (5.848) | 49.60 (3.857) | 67.859 (9.4141)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 173.00 (5.657) | 161.00 (4.243) | 166.50 (6.364) | 162.8 (7.85) | 167.0 (NA) — Standard deviation was not estimable since only one participant was analyzed. | 164.7 (6.47) | 163.0 (8.15) | 172.3 (7.23) | 154.7 (2.52) | 164.09 (7.485)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 23.90 (4.808) | 26.23 (2.636) | 23.75 (3.182) | 26.62 (1.599) | 24.30 (NA) — Standard deviation was not estimable since only one participant was analyzed. | 24.53 (1.401) | 26.42 (2.872) | 26.47 (3.202) | 20.77 (1.553) | 25.16 (2.775)

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Number of Participants Who Experienced at Least One Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Event (SAE)
Time Frame: Baseline up to Day 60
Population: The safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Non-Japanese Cohort 1; Period A: Placebo: TAK-418 placebo-matching capsule, orally, once on Day 1 of Period A.
- Non-Japanese Cohort 1; Period B: Placebo: TAK-418 placebo-matching capsule, orally, once on Day 1 of Period B.
- Non-Japanese Cohort 1: TAK 418 120 mg: TAK-418 120 mg, capsule, orally, once on Day 1 of Period A.
- Non-Japanese Cohort 1: TAK 418 160 mg: TAK-418 160 mg, capsule, orally, once on Day 1 of Period B.
Arm/Group | Non-Japanese Cohort 1; Period A: Placebo | Non-Japanese Cohort 1; Period B: Placebo | Non-Japanese Cohort 1: TAK 418 120 mg | Non-Japanese Cohort 1: TAK 418 160 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Participants
  TEAE | 1 | 0 | 3 | 2
  SAE | 0 | 0 | 0 | 0

2. Primary Outcome: Cohorts 2 to 5: Number of Participants Who Experienced at Least One TEAEs and SAE
Time Frame: Baseline up to Day 70
Population: The safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Japanese Cohorts 2 to 4: Pooled Placebo | Japanese Cohort 5: Placebo | Non-Japanese Cohort 2: TAK-418 20 mg | Non-Japanese Cohort 3: TAK-418 60 mg | Non-Japanese Cohort 4: TAK-418 160 mg | Japanese Cohort 5: TAK-418 20 mg
Number analyzed (Participants) | 5 | 1 | 6 | 6 | 3 | 3
Participants
  TEAE | 3 | 1 | 5 | 6 | 3 | 1
  SAE | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Cohort 1: Number of Participants With Markedly Abnormal Criteria for Clinical Laboratory Values at Least Once Postdose
Time Frame: Baseline up to Day 60
Population: The safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Japanese Cohort 1; Period A: Placebo | Non-Japanese Cohort 1; Period B: Placebo | Non-Japanese Cohort 1: TAK 418 120 mg | Non-Japanese Cohort 1: TAK 418 160 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Participants | 0 | 0 | 0 | 1

4. Primary Outcome: Cohorts 2 to 5: Number of Participants With Markedly Abnormal Criteria for Clinical Laboratory Values at Least Once Postdose
Time Frame: Baseline up to Day 70
Population: The safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Japanese Cohorts 2 to 4: Pooled Placebo | Japanese Cohort 5: Placebo | Non-Japanese Cohort 2: TAK-418 20 mg | Non-Japanese Cohort 3: TAK-418 60 mg | Non-Japanese Cohort 4: TAK-418 160 mg | Japanese Cohort 5: TAK-418 20 mg
Number analyzed (Participants) | 5 | 1 | 6 | 6 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Cohort 1: Number of Participants With Markedly Abnormal Criteria for Vital Signs at Least Once Postdose
Time Frame: Baseline up to Day 60
Population: The safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Japanese Cohort 1; Period A: Placebo | Non-Japanese Cohort 1; Period B: Placebo | Non-Japanese Cohort 1: TAK 418 120 mg | Non-Japanese Cohort 1: TAK 418 160 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Participants
  Pulse Rate less than (<) 50 beats per minute (bpm) | 0 | 1 | 1 | 0
  Systolic Blood Pressure <85 mmHg | 0 | 0 | 0 | 1
  Temperature <35.6 Celsius (C) | 0 | 1 | 1 | 1

6. Primary Outcome: Cohorts 2 to 5: Number of Participants With Markedly Abnormal Criteria for Vital Signs at Least Once Postdose
Time Frame: Baseline up to Day 70
Population: The safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Japanese Cohorts 2 to 4: Pooled Placebo | Japanese Cohort 5: Placebo | Non-Japanese Cohort 2: TAK-418 20 mg | Non-Japanese Cohort 3: TAK-418 60 mg | Non-Japanese Cohort 4: TAK-418 160 mg | Japanese Cohort 5: TAK-418 20 mg
Number analyzed (Participants) | 5 | 1 | 6 | 6 | 3 | 3
Participants
  Diastolic Blood Pressure <50 mmHg | 0 | 0 | 0 | 2 | 0 | 0
  Pulse Rate greater than (>) 120 bpm | 1 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure <85 mmHg | 0 | 0 | 0 | 0 | 0 | 1

7. Primary Outcome: Cohort 1: Number of Participants Who Meet the Markedly Abnormal Values of 12-lead Electrocardiogram (ECG) Parameters at Least Once Post Dose
Time Frame: Baseline up to Day 60
Population: The safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Japanese Cohort 1; Period A: Placebo | Non-Japanese Cohort 1; Period B: Placebo | Non-Japanese Cohort 1: TAK 418 120 mg | Non-Japanese Cohort 1: TAK 418 160 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Participants
  ECG Mean Heart Rate <50 bpm | 0 | 1 | 0 | 1
  QT Interval >=460 millisecond (msec) | 0 | 0 | 1 | 0

8. Primary Outcome: Cohorts 2 to 5: Number of Participants Who Meet the Markedly Abnormal Values of 12-lead ECG Parameters at Least Once Post Dose
Time Frame: Baseline up to Day 70
Population: The safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Japanese Cohorts 2 to 4: Pooled Placebo | Japanese Cohort 5: Placebo | Non-Japanese Cohort 2: TAK-418 20 mg | Non-Japanese Cohort 3: TAK-418 60 mg | Non-Japanese Cohort 4: TAK-418 160 mg | Japanese Cohort 5: TAK-418 20 mg
Number analyzed (Participants) | 5 | 1 | 6 | 6 | 3 | 3
Participants | 1 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Cohort 1; AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-418 on Day 1
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The pharmacokinetic (PK) set included all participants from the safety set who had at least 1 measurable post dose plasma or cerebrospinal fluid (CSF) concentration or amount of drug in urine of TAK-418F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Non-Japanese Cohort 1: TAK 418 120 mg | Non-Japanese Cohort 1: TAK 418 160 mg
Number analyzed (Participants) | 6 | 6
hour*nanogram per milliliter (hr*ng/mL) | 3761.2 (20.8) | 4229.0 (40.4)

10. Secondary Outcome: Cohort 2 to 5: AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Over the Dosing Interval for TAK-418 on Days 1 and 10
Time Frame: Days 1 and 10 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: The PK set included all participants from the safety set who had at least 1 measurable post dose plasma or CSF concentration or amount of drug in urine of TAK-418F.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Non-Japanese Cohort 2: TAK-418 20 mg | Non-Japanese Cohort 3: TAK-418 60 mg | Non-Japanese Cohort 4: TAK-418 160 mg | Japanese Cohort 5: TAK-418 20 mg
Number analyzed (Participants) | 6 | 6 | 3 | 3
hr*ng/mL
  Day 1 | 503.3 (165.71) | 1445.5 (353.26) | 3747.3 (239.53) | 610.3 (87.89)
  Day 10 | 668.2 (228.83) | 1660.5 (421.77) | 4058.3 (249.49) | 677.3 (73.66)

11. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-418
Time Frame: Cohort 1: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose; Cohorts 2 to 5: Days 1 and 10 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The PK set included all participants from the safety set who had at least 1 measurable post dose plasma or CSF concentration or amount of drug in urine of TAK-418F. PK-evaluable population where data at specified time points was available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Non-Japanese Cohort 1: TAK 418 120 mg | Non-Japanese Cohort 1: TAK 418 160 mg | Non-Japanese Cohort 2: TAK-418 20 mg | Non-Japanese Cohort 3: TAK-418 60 mg | Non-Japanese Cohort 4: TAK-418 160 mg | Japanese Cohort 5: TAK-418 20 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 3
nanogram per milliliter (ng/mL)
  Day 1 | 714.7 (21.6) | 750.3 (40.3) | 81.1 (35.8) | 270.8 (21.6) | 657.8 (33.0) | 154.5 (5.9)
  Day 10: number analyzed (Participants) | 0 | 0 | 6 | 6 | 3 | 3
  Day 10 |  |  | 113.4 (30.8) | 303.4 (17.6) | 692.4 (15.4) | 171.1 (5.9)

12. Secondary Outcome: Tmax: Time to Reach the Cmax for TAK-418
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Median (Full Range); unit: hour
Arm/Group | Non-Japanese Cohort 1: TAK 418 120 mg | Non-Japanese Cohort 1: TAK 418 160 mg | Non-Japanese Cohort 2: TAK-418 20 mg | Non-Japanese Cohort 3: TAK-418 60 mg | Non-Japanese Cohort 4: TAK-418 160 mg | Japanese Cohort 5: TAK-418 20 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 3
hour
  Day 1 | 1.500 [1.00 to 1.50] | 1.250 [1.00 to 2.00] | 1.750 [1.00 to 3.00] | 1.500 [1.00 to 4.00] | 1.500 [1.00 to 3.00] | 1.000 [0.50 to 1.50]
  Day 10: number analyzed (Participants) | 0 | 0 | 6 | 6 | 3 | 3
  Day 10 |  |  | 1.260 [1.00 to 2.00] | 1.250 [1.00 to 3.00] | 1.000 [1.00 to 1.50] | 1.000 [1.00 to 1.50]

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events (AEs) that started after the first dose of study drug and no more than 30 days after the last dose of study drug (up to Day 60 in Cohort 1 and Day 70 in Cohorts 2 to 5)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Non-Japanese Cohort 1; Period A: Placebo | Non-Japanese Cohort 1; Period B: Placebo | Non-Japanese Cohort 1: TAK 418 120 mg | Non-Japanese Cohort 1: TAK 418 160 mg | Non-Japanese Cohorts 2 to 4: Pooled Placebo | Japanese Cohort 5: Placebo | Non-Japanese Cohort 2: TAK-418 20 mg | Non-Japanese Cohort 3: TAK-418 60 mg | Non-Japanese Cohort 4: TAK-418 160 mg | Japanese Cohort 5: TAK-418 20 mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/6 | 0/6 | 0/5 | 0/1 | 0/6 | 0/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/6 | 0/6 | 0/5 | 0/1 | 0/6 | 0/6 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/2 | 0/2 | 3/6 | 2/6 | 3/5 | 1/1 | 5/6 | 6/6 | 3/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Japanese Cohort 1; Period A: Placebo (N=2) | Non-Japanese Cohort 1; Period B: Placebo (N=2) | Non-Japanese Cohort 1: TAK 418 120 mg (N=6) | Non-Japanese Cohort 1: TAK 418 160 mg (N=6) | Non-Japanese Cohorts 2 to 4: Pooled Placebo (N=5) | Japanese Cohort 5: Placebo (N=1) | Non-Japanese Cohort 2: TAK-418 20 mg (N=6) | Non-Japanese Cohort 3: TAK-418 60 mg (N=6) | Non-Japanese Cohort 4: TAK-418 160 mg (N=3) | Japanese Cohort 5: TAK-418 20 mg (N=3)
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 4 | 5 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Food aversion (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypervigilance (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT03501069/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT03501069/SAP_001.pdf